CLINICAL TRIAL: NCT05475691
Title: Protocol-LATAM RegistrAME: Longitudinal Data Collection in Pediatric and Adult Patients With Spinal Muscular Atrophy in Latin America - a Regional Registry
Brief Title: Longitudinal Data Collection in Pediatric and Adult Patients With Spinal Muscular Atrophy in Latin America
Acronym: RegistrAME
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Otavio Berwanger, Director ARO (Academic Research Organization), Hospital Israelita Albert Einstein
Other Study IDs: Protocol-LATAM RegistrAME
Record Dates: First submitted 2022-07-19; First posted 2022-07-27 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy 1; Spinal Muscular Atrophy 2; Spinal Muscular Atrophy 3; Spinal Muscular Atrophy 4; SMN1 gene; Nusinersen; onasemnogene abeparvovec; Small molecule drug
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood; Spinal muscular atrophy 4; Spinal Muscular Atrophy, Type IV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Type 1 SMA (with and without use of disease-modifying treatment (DMTs)): * Participants of both sexes who presented signs and symptoms of Spinal Muscular Atrophy before six months of age and have a genetic report confirming 5q SMA.
  * No interventions will be performed in this study (RegistrAME is observational study (retrospective and prospective) non-randomized, international multicenter study- Registration of patients in Latin America).
  * Data collection aims to gather as much information as possible regarding the clinical profile of patients, interventions performed in the routine of care and clinical evolution over time (Real World Evidence-RWE).
  * The planned SMA registry will provide an online platform to collect longitudinal data on SMA patients across Latin America to achieve a better understanding of the clinical characteristics of SMA patients, the natural history of the disease and the use of DMTs (on participants who are using DMTs).
- Type 2 SMA (with and without disease-modifying treatment (DMTs)): * Participants of both sexes who presented signs and symptoms of Spinal Muscular Atrophy starting between six and eighteen months of age and have a genetic report confirming 5q SMA.
  * No interventions will be performed in this study (RegistrAME is observational study (retrospective and prospective) non-randomized, international multicenter study- Registration of patients in Latin America).
  * Data collection aims to gather as much information as possible regarding the clinical profile of patients, interventions performed in the routine of care and clinical evolution over time (Real World Evidence-RWE).
  * The planned SMA registry will provide an online platform to collect longitudinal data on SMA patients across Latin America to achieve a better understanding of the clinical characteristics of SMA patients, the natural history of the disease and the use of DMTs (on participants who are using DMTs).
- Type 3 SMA (with and without disease-modifying treatment (DMTs)): * Participants of both sexes who presented the first signs and symptoms of Spinal Muscular Atrophy starting after eighteen months of age and have a genetic report confirming 5q SMA.
  * No interventions will be performed in this study (RegistrAME is observational study (retrospective and prospective) non-randomized, international multicenter study- Registration of patients in Latin America).
  * Data collection aims to gather as much information as possible regarding the clinical profile of patients, interventions performed in the routine of care and clinical evolution over time (Real World Evidence-RWE).
  * The planned SMA registry will provide an online platform to collect longitudinal data on SMA patients across Latin America to achieve a better understanding of the clinical characteristics of SMA patients, the natural history of the disease and the use of DMTs (on participants who are using DMTs).
- Type 4 SMA (with and without disease-modifying treatment (DMTs)): * Participants of both sexes and that the first symptoms of Spinal Muscular Atrophy appeared from the second or third decade of life and have a genetic report confirming 5q SMA.
  * No interventions will be performed in this study (RegistrAME is observational study (retrospective and prospective) non-randomized, international multicenter study- Registration of patients in Latin America).
  * Data collection aims to gather as much information as possible regarding the clinical profile of patients, interventions performed in the routine of care and clinical evolution over time (Real World Evidence-RWE).
  * The planned SMA registry will provide an online platform to collect longitudinal data on SMA patients across Latin America to achieve a better understanding of the clinical characteristics of SMA patients, the natural history of the disease and the use of DMTs (on participants who are using DMTs).

SUMMARY:
The natural history of SMA patients has changed, due to the improvements in treatment and technological advances. The systematic collection of data from routine clinical practice in multiple Latin American countries, harmonized to an internationally aligned core data set, is important to advancing the understanding the natural history of disease in the region and the influence of different drug treatments on patient outcomes. These data are critical to improving the care of these patients. So far, clinical trials regarding therapeutic approaches for SMA patients only cover a subgroup of the broad spectrum of severity of SMA. Thus, there is a strong need to monitor the full range of treated and untreated SMA patients in a real-world context.The aim of this study is to set up a regional healthcare provider (HCP) entered registry. The planned SMA registry will provide an online platform to collect longitudinal data on SMA patients across Latin America to achieve a better understanding of the clinical characteristics of SMA patients, the natural history of the disease, the use of DMTs and patients' outcomes, as well as to support further research projects and regional data generation.

DETAILED DESCRIPTION:
This is a retrospective and prospective, multicenter non-randomized registry in Latin America. The variables included in the RegistrAME registry are based on the core items defined by the TREAT-NMD for SMA registries and the RegistrAME steering committee consensus. Items such as demographic characteristics, date of genetic test result, clinical diagnosis, functional status and pulmonary function, among others, are included in RegistrAME. The RegistrAME registry will allow the inclusion of retrospective clinical data in those centers where natural history studies of for spinal muscular atrophy are currently being conducted. RegistrAME will also offer a standardized structure for prospective data collection in all centers. The current aim of this registry is to include centres in LATAM meeting the structural and personnel requirements for performing the planned regular registry-related investigations. These reference centers in LATAM (Latin America) will be selected from COEs which 1) have the potential to enroll and make the proper patient follow up, 2) have experience in treating SMA, and 3) have experience in conducting clinical trials. An electronic Case Report Form (e-CRF) will be created by the ARO (Academic Research Organization) from Hospital Albert Einstein, using REDCap (Research Electronic Data Capture). The electronic Case Report Form (e-CRF) created to meet international standards for data protection and quality management, and to harmonize the platform with those currently used by other countries. No interventions will be performed in this study, the RegistrAME is observational study non-randomized, international multicenter study (Registration of patients in Latin America). Data collection aims to gather as much information as possible regarding the clinical profile of patients, interventions performed in the routine of care and clinical evolution over time (Real World Evidence-RWE). After confirmation of eligibility and informed consent, patients will undergo medical evaluation, and then retrospective data collection (when possible and limited to 6 months before the patient inclusion in the study), baseline data and continuation of longitudinal data collection will be started. Data entry is planned to be performed every carried out at intervals of 4 to 6 months (according to the type of SMA), depending on the regular healthcare planning of each clinical site. The study will assess disease progression, both the natural history of the disease and the effectiveness of different SMA specific drug treatments on patient outcomes. Duration of disease, survival with or without ventilatory support, motor function, pulmonary function, developmental milestones achieved, growth parameters, orthopedic symptoms, functional assessments (CHOP-INTEND (Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders), HINE-2 (Hammersmith Infant Neuromuscular Examination - session 2), HFMSE (Hammersmith Motor Functional Scale Expanded), RULM (Revised Upper Limb Module), and 6MWT (The six minute walking test)) will be analyzed depending on the functional capacity of the patients and 5q SMA type over time.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed 5q SMA patients at all ages;
* Consent to participate in the study, expressed by the patient or responsible or legal guardian of the pediatric patient/ responsible or legal guardian of the patient with cognitive impairment of understanding the registration protocol.

Exclusion Criteria:

* Patients without a genetic diagnosis confirming SMA 5q;
* Other types of SMA (non 5q SMA);
* Patients who do not accept to participate in the observational study;
* Patients without the legal capacity who are unable to understand the nature, significance and consequences of participating in the registry, or, in such cases, without a legal or responsible guardian.

Min Age: 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with SMA 5q Types 1, 2, 3 and 4 (with and without disease-modifying treatment) of all ages and both sexes.
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Describe the natural history of the disease (5q SMA in patients in Latin America) in a real-life context. | 24 months (Study duration time)
  Characterization and description the evolution of the patient's condition over the time of data collection from the registry, to describe the natural history of the disease in a real-life context.

SECONDARY OUTCOMES:
Disease characteristics at first diagnosis. | Baseline
  Early signs and symptoms leading to clinical diagnosis of SMA

OTHER OUTCOMES:
Duration of disease. | 24 months (Study duration time)
  Time interval between the age of appearance of the first signs and symptoms to the current age
Time from SMA symptom onset until genetic diagnosis. | Baseline
  To verify heterogeneity of access resources to genetic diagnosis.
Motor milestones over time. | 24 months
  Motor functions (unable to sit, sitting without support, walking with support; standing without Support; walking independently) will be evaluated over time.
Expanded Hammersmith Functional Motor Scale | 24 months
  Hammersmith Functional Motor Scale-Expanded (HFMSE) scores range from 0 to 66,
Revised Upper Limb Module | 24 months
  Revised Upper Limb Module (RULM) scores range from 0 to 37, with higher scores indicating better function.
Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders Scale (CHOP-INTEND) | 24 months
  CHOP-INTEND (Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders) scores range from 0 to 64 with higher scores indicating better function.
Gain and loss of motor function | 24 months (Study duration time)
  Analyze throughout the study "Shift up (gained motor function)", "No change" and "Shift down" (loss of motor function) over time, in the different types of 5qSMA with and without disease-modifying treatment.
History of hospitalizations | 24 months (Study duration time)
  Records of need for hospitalizations
History and characterization of previous surgical procedures and need for surgery | 24 months (Study duration time)
  History of comorbidities
Utilization of DMTs - Disease Modifying Treatments | 24 months (Study duration time)
  History of use or non-use of DMTs
Use of Medications | 24 months (Study duration time)
  Analysis of the history of drugs used in the clinical routine of patients
Pulmonary Function | 24 months (Study duration time)
  Frequency and length of time of ventilatory support use

CONTACTS AND LOCATIONS:
Overall Officials: Otávio Berwanger, PhD, Study Director — Hospital Albert Einstein; Henrique Fonseca, PhD, Study Director — Hospital Albert Einstein
Locations (18):
- Argentina (5):
  - Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires F.D.
  - Hospital de Pediatria J.P.Garrahan, Buenos Aires, Buenos Aires F.D.
  - Private office, Buenos Aires, Rivadavia 4951 PB 2 Caballito
  - Clínica Universitaaria Reina Fabiola, Córdoba
  - Hospital Pediátrico Humberto Notti, Mendoza
- Brazil (8):
  - HUPES - Escola Bahiana de Medicina e Saúde Pública, Salvador, Estado de Bahia
  - UFMG - Universidade Federal de Minas Gerais - Hospital das Clínicas, Belo Horizonte, Minas Gerais
  - Hospital Infantil Pequeno Príncipe, Curitiba, Paraná
  - Instituto de Puericultura e Pediatria Martagão Gesteira da UFRJ, Rio de Janeiro, Rio de Janeiro
  - HCPA - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Unicamp - Hospital de Clínicas da Universidade Estadual de Campinas, Campinas, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
  - Instituto da Criança do Hospital das Clínicas de São Paulo - FMUSP, São Paulo, São Paulo
- Clínica Meds La Dehesa, Santiago, Chile
- Colombia (2):
  - Fundação Hospital da Misericórdia, Bogotá
  - Instituto Roosevelt Pontifícia Universidade Javeriana, Bogotá
- Hospital Christus Muguerza Alta Especialidade, Monterrey, Mexico
- Centro Hospitalario Pereira Rossell, Facultad de Medicina- Universidad de la Republica, Montevideo, Uruguay

REFERENCES:
- [Derived] Batista EC, Zanoteli E, Monfardini F, Santos GPD, Silva GS, Berwanger O, Rizzo LV, Fonseca HARD. Longitudinal data collection in pediatric and adult patients with 5q spinal muscular atrophy in Latin America: LATAM RegistrAME study - a clinical registry study protocol. Einstein (Sao Paulo). 2024 Dec 9;22:eAE1133. doi: 10.31744/einstein_journal/2024AE1133. eCollection 2024. PMID 39661851